CLINICAL TRIAL: NCT05410912
Title: Varicose Vein in Patients Under the Age of 40
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Ziheng Wu, MD, Associated chief physician, First Affiliated Hospital of Zhejiang University
Other Study IDs: IIT20210662A
Record Dates: First submitted 2022-06-06; First posted 2022-06-08 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- The younger group: Patients who were under the age of 40
  Interventions: Procedure: Great saphenous vein stripping and ambulatory phlebectomy
- The older group: Patients who were more than 40 years old
  Interventions: Procedure: Great saphenous vein stripping and ambulatory phlebectomy

INTERVENTIONS:
Procedure: Great saphenous vein stripping and ambulatory phlebectomy — All patients included in the study were treated with great saphenous vein stripping and ambulatory phlebectomy.

SUMMARY:
Varicose veins are a result of valvular insufficiency and presented with twisted, enlarged veins. They not only cause cosmetic concerns but also lead to limb edema, skin pigmentation/lipodermatosclerosis, and even venous ulcers. This disease affects a large percentage of the population. Although there have been several researches on the risk factors for varicose veins and the outcomes of alternative therapies , there is currently limited data focusing on varicose veins in young patients. In this case-control study, we wanted to assess the risk factors for varicose veins in patients under the age of 40, as well as their long-term results of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. great saphenous varicose veins (GSVV) with saphenous vein reflux >0.5s.
2. lower extremity venography excluding iliac vein compression;
3. treated by great saphenous vein stripping and ambulatory phlebectomy.
4. the patient had a minimum follow-up of five years.

Exclusion Criteria:

1. secondary varicose veins (defined as varicose veins caused by deep vein thrombosis, iliac venous compression or venous injury etc.);
2. small saphenous veins;
3. treated by endovenous ablation/laser or sclerotherapy alone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary great saphenous varicose veins (GSVV) and treated by great saphenous vein stripping and ambulatory phlebectomy.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative varicose veins sequelae | Five years after surgery.
  The sequelae of the varicose vein were assessed by Venous Clinical Severity Score (VCSS). The total score is 0~30. The higher scores mean a worse outcome.
Postoperative quality of life | Five years after surgery.
  Quality of life was assessed by the Aberdeen Varicose Vein Questionnaire (AVVQ). The total score is 1~100. The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided